CLINICAL TRIAL: NCT00701857
Title: Phase I Study of Concomitant Pemetrexed and CDDP Plus Radiation Therapy in Patients With Locally Advanced or Metastatic Esophageal or Gastroesophageal (GEJ) Carcinomas
Brief Title: Pemetrexed, Cisplatin, and Radiation Therapy in Treating Patients With Esophageal or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0612-04; P30CA023074 (NIH); UARIZ-07-0612-04 (Other: University of Arizona); UARIZ-BIO07067 (Other: University of Arizona); UARIZ-SRC18084 (Other: University of Arizona); LILLY-UARIZ-07-0612-04 (Other Grant/Funding Number: Eli Lilly)
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Esophageal Cancer
Keywords: stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin; Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed, Cisplatin, Radiation Therapy (Experimental): Concomitant Pemetrexed and CDDP Plus Radiation Therapy
  Interventions: Drug: cisplatin; Drug: Pemetrexed; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Standard weekly dose
  Other Names: CDDP
Drug: Pemetrexed — Biweekly pemetrexed dose escalation
  Other Names: Pemetrexed disodium
Radiation: radiation therapy — Weekly standard dose radiation therapy
  Other Names: RT

SUMMARY:
RATIONALE: Pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Cisplatin may make tumor cells more sensitive to radiation therapy. Giving pemetrexed together with cisplatin and radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of pemetrexed when given together with cisplatin and radiation therapy in treating patients with stage III or stage IV esophageal cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the maximum tolerated dose of pemetrexed disodium in combination with cisplatin and standard-dose radiotherapy in patients with stage III or IV esophageal or gastroesophageal junction carcinoma.

Secondary

* To specifically characterize the toxicity profile of this regimen.
* To investigate, preliminarily, the anti-tumor activity of this regimen, as measured by standard response criteria (RECIST criteria), in patients with measurable disease.

OUTLINE: This is a dose-escalation study of pemetrexed disodium.

Patients receive pemetrexed disodium IV over 10 minutes on days 1, 15, and 29 and cisplatin IV over 10 minutes on days 1, 8, 15, 22, and 29. Patients also undergo external beam radiotherapy once daily, 5 days a week, for up to 6 weeks.

After completion of study therapy, patients are followed for 30 days and then every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of esophageal or gastroesophageal junction carcinoma

  * Stage III or IV disease
* Treatment with chemoradiotherapy is considered appropriate
* Measurable or evaluable disease
* Clinically significant pleural or pericardial effusions or ascites allowed provided they were drained prior to study entry

  * No pleurodesis within the past 2 weeks
* Controlled brain metastasis allowed provided patient is clinically stable with no signs of progression by MRI or CT scan of the brain ≥ 60 days after completion of treatment AND is asymptomatic and does not require steroids

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* WBC ≥ 2,500/mm^3
* ANC ≥ 1,500/mm^3
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm^3
* Total bilirubin normal
* Alkaline phosphatase AND AST and ALT meeting the following criteria:

  * Alkaline phosphatase normal AND AST or ALT ≤ 3 times upper limit of normal (ULN) (≤ 5 times ULN for patients with liver metastases)
  * Alkaline phosphatase ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * Alkaline phosphatase ≤ 5 times ULN AND AST or ALT normal
* Creatinine clearance ≥ 45 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* Able to take folic acid, vitamin B_12, or corticosteroids
* No known severe hypersensitivity reaction to study drugs
* No uncontrolled serious active infection
* No pre-existing peripheral neuropathy > grade 1
* No significant cardiac disease, including any of the following:

  * Uncontrolled high blood pressure
  * Unstable angina
  * Congestive heart failure within the past 6 months
  * Left ventricular ejection fraction below the lower limit of normal
  * Myocardial infarction within the past year
  * Serious cardiac arrhythmias requiring medication

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic therapy regimens
* No prior radiotherapy to gastric/esophageal fields
* No aspirin or other NSAID before and after pemetrexed disodium administration
* No concurrent colony-stimulating factors (CSF) to maintain WBC and ANC eligibility values

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2014-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of pemetrexed | 6 months

SECONDARY OUTCOMES:
Toxicity profile | 12 months
Response (complete response, partial response, progressive disease, and stable disease) as measured by RECIST criteria | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Emad Elquza, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

REFERENCES:
- [Derived] Elquza E, Babiker HM, Howell KJ, Kovoor AI, Brown TD, Patel H, Malangone SA, Borad MJ, Dragovich T. Phase I Study of Concomitant Pemetrexed and Cisplatin Plus External Beam Radiation Therapy in Patients with Locally Advanced or Metastatic Esophageal or Gastroesophageal Junction Carcinomas. Cancer Invest. 2016;34(2):57-63. doi: 10.3109/07357907.2015.1108426. Epub 2016 Jan 25. PMID 26810581